CLINICAL TRIAL: NCT01612039
Title: A Phase 2, Randomized, Double-Blind, Parallel, Placebo-Controlled, Proof-of-Concept Study to Assess the Efficacy, Safety, and Tolerability of ASP3291 in Patients With Active Ulcerative Colitis
Brief Title: Safety, Efficacy, and Tolerability Study of ASP3291 in Patients With Active Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Telsar Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3291-CL-0004
Record Dates: First submitted 2012-06-01; First posted 2012-06-05 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Ulcerative Colitis
Keywords: ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ASP3291 (Experimental)
  Interventions: Drug: ASP3291
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP3291 — Tablet, 1,000 mg (four 250-mg tablets), twice a day, 8 weeks
  Arms: ASP3291
Drug: Placebo — Matching placebo tablets
  Arms: Placebo

SUMMARY:
This is a Phase 2, randomized, double-blind, multicenter, parallel, placebo controlled study. Approximately 120 eligible patients with mild-to-moderate active ulcerative colitis will be randomized to double blind treatment of either 1,000 mg twice daily (b.i.d.) ASP3291 (2,000 mg/d) or matching placebo in a 1:1 ratio for 8 weeks.

The study hypothesis is that treatment with ASP3291 compared to placebo will improve a patient's ulcerative colitis endoscopic score from baseline to Week 8.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of ulcerative colitis by endoscopy and histology consistent with diagnosis
* Must be able to provide informed consent
* Has a Modified Baron Score of at least 2 (as determined by the investigator) at 15 cm or more from the anal verge as assessed during the screening period
* Has an Ulcerative Colitis Clinical Score (UCCS) of at least 4, with a stool frequency and rectal bleeding score of at least 1 as assessed during the screening period
* If female, is at least 2 years postmenopausal, surgically sterile per documentation provided by a medical professional, agrees to sexual abstinence, or uses two approved highly effective methods of birth control during the study period and for 30 days after the last dose of study drug
* If male, agrees to sexual abstinence or to use two highly effective methods of birth control during the study period and for 90 days after last dose; agrees to not donate sperm during the study period and for 90 days after last dose
* Willing and able to comply with the study requirements

Exclusion Criteria:

* Has a history of any clinically significant neurological, renal, hepatic, gastrointestinal, pulmonary, metabolic, cardiovascular, psychiatric, endocrine, hematological disorder or disease, or any other medical condition that, in the investigator's opinion, would preclude participation in the study
* Has severe Ulcerative Colitis as defined by an average bloody stool frequency of >6 per day and at least one of the following:

  * Resting heart rate >90 bpm
  * Oral temperature of >38°C (>100.4°F)
  * Hemoglobin of <10.5 g/dL
* Has has undergone previous resective colonic surgery
* Has a significant or immediate risk for toxic megacolon
* Has previous diagnosis with Crohn's disease, indeterminate colitis, microscopic colitis or acute diverticulitis based on medical history
* Has an extension of disease limited to ulcerative proctitis (i.e., disease extension less than 15 cm from the anal verge)
* Has an active peptic ulcer disease based on medical history
* Shows a stool culture positive for enteric pathogens during the screening period
* Had previous treatment with tumor necrosis factor-α (TNF α) inhibitors
* Had treatment with rectal corticosteroid within 2 weeks before Day -2
* Has active liver disease or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2 times the upper limit of normal (ULN) at screening
* Has an estimated glomerular filtration rate (using Cockroft-Gault formula corrected for body surface area) of <60 mL/min at screening
* Known history of human immunodeficiency virus antibody
* History of severe allergic or anaphylactic reactions requiring medical attention
* Has participated in another investigational study within 30 days before Visit 3
* History of drug or alcohol abuse in the past 2 years
* Has previously participated in a study with ASP3291

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2012-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline (Visit 2) to Week 8 (Visit 7) in Modified Baron Score | Baseline to Week 8

SECONDARY OUTCOMES:
Proportion of subjects with Modified Baron Score of 0 or 1 at Week 8 (Visit 7) | Week 8
Change in Ulcerative Colitis Clinical Score of >3 | Basline to Week 8
Ulcerative Colitis Clinical Score stool frequency and rectal bleeding score of 0 | Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Robert Schinagl, Ph.D., Study Director — Drais Pharmaceuticals, Inc.

IPD SHARING:
Plan to Share IPD: No